CLINICAL TRIAL: NCT04348383
Title: Phase IIb Prospective, Multi-center, Randomized, Parallel, Double Blind, Placebo Controlled Trial to Evaluate Defibrotide Intravenous Infusion in the Prevention and Treatment of COVID-19 Respiratory Distress and Cytokine Release Syndrome
Brief Title: Defibrotide as Prevention and Treatment of Respiratory Distress and Cytokine Release Syndrome of Covid 19.
Acronym: DEFACOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMIB-DFC-2020-02
Record Dates: First submitted 2020-04-08; First posted 2020-04-16 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2022-06

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — defibrotide

STUDY DESIGN:
Intervention Model Description: Phase IIb prospective, multi-center, randomized, parallel, double blind, placebo controlled
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Defibrotide + standard therapy (Experimental): Defibrotide + standard therapy
  Interventions: Drug: Defibrotide
- Placebo (Placebo Comparator): Placebo + standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Defibrotide — 6.25 mg/kg every 6 hours in 2 hours infusion for 7 or 15 days
  Arms: Defibrotide + standard therapy
Drug: Placebo — Placebo 250 cc every 6 hours for 7 or15 days
  Arms: Placebo

SUMMARY:
Protection of endothelial dysfunction by intravenous infusion of Defibrotide (Defitelio), expected to decrease inflammation and expression of adhesion molecules in the endothelium, leukocyte tissue infiltration and epithelial destruction, and to promote immune tolerance through a change in the Cytokine balance, which is decisive in preventing multiorgan failure and death in patients with SARS-CoV-2 infection with clinical status grade 4 or 5 according to the WHO classification

DETAILED DESCRIPTION:
Protection of endothelial dysfunction by intravenous infusion of Defibrotide (Defitelio), expected to decrease inflammation and expression of adhesion molecules in the endothelium, leukocyte tissue infiltration and epithelial destruction, and to promote immune tolerance through a change in the Cytokine balance, which is decisive in preventing multiorgan failure and death in patients with SARS-CoV-2 infection with clinical status grade 4 or 5 according to the WHO classification

ELIGIBILITY:
Inclusion Criteria:

1. Acceptance of participation in the study by the patient or legal representative.
2. Patients of any gender, 18 years or older.
3. Confirmed diagnosis by PCR+ of SARS-CoV-2 infection.
4. COVID-19 positive patients WHO grades 4, 5 or 6.

   * Grade 4: hospitalized requiring oxygen therapy.
   * Grade 5: hospitalized requiring high-flow oxygen therapy, noninvasive mechanical ventilation, or both.
5. Levels of IL-6 ≥ 3 times the upper limit of normality

Exclusion Criteria:

1. Acute bleeding.
2. Thrombolytic treatment and anticoagulant treatment at therapeutic doses.
3. Pregnancy or lactation.
4. Patients with active malignant tumour, other serious systemic or neuropsychiatric diseases.
5. Patients participating in other clinical trials in the last month.
6. Inability to give informed consent or to accomplish the requirements of the diagnostic tests.
7. Patients with hypersensitivity to Defibrotide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Clinical improvement. | 7,15, 30 day
  Number of days that the patient maintains the clinical improvement. The patient achieves a change of al least 1 category on WHO scale.

SECONDARY OUTCOMES:
1. Mortality rate | : up to 30 days
  All cause mortality
Rate os serious adverse events . | 7, 15, 30 and 60 Day
  Number of adverse events with possible, probable or definite relationship with the study.
Clinical improvement by WHO | 7, 15, 30 and 60 Day
  Decrease ventilation days in grade 6 patients
Clinical improvement by NEWS2 scales | 7, 15, 30 and 60 Day
  Decrease the rate of grades 4-5 patients requiring mechanical ventilation.
Clinical improvement by NEWS2 scales | 7, 15, 30 and 60 Day
  Decrease ventilation days in grade 6 patients
Biologic response | 7, 15, 30 and 60 Day
  Decrease of IL-6 levels with respect to the basal ones > 50%.
Biologic response | 7, 15, 30 and 60 Day
  Absolute lymphocytes count: 50% increase with respect to the baseline
Biologic response | 7, 15, 30 and 60 Day
  Normal D-dimer (DD) or decrease of 50% with respect to the baseline
Biologic response | 7, 15, 30 and 60 Day
  Normal CRP or decrease of 50% with respect to the baseline
Biologic response | 7, 15, 30 and 60 Day
  Normal LDH or decrease of 50% with respect to the baseline
Biologic response | 7, 15, 30 and 60 Day
  Normal CPK or decrease of 50% with respect to the baseline
Biologic response | 7, 15, 30 and 60 Day
  Normal Ferritin or decrease of 50% with respect to the baseline
Radiological response | 7, 15, 30 and 60 Day
  Improvement of radiological images by conventional radiology
Collection and storage of biological samples | 15,30 days
  improve the knowledge of the disease at the inclusion of the patients
Clinical improvement by WHO | 7, 15, 30 and 60 Day
  Decrease the rate of grades 4-5 patients requiring mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Clinico y Provincial de Barcelona, Barcelona
  - Virgen de la Arrixaca University Clinical Hospital, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital General Universitario Reina Sofía, Murcia
  - Hospital Universitario Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No